CLINICAL TRIAL: NCT05699915
Title: Extensive CArdioVAscular Characterization and Follow-up of Patients Receiving Immune Checkpoint Inhibitors: a Prospective Multicentre Study
Brief Title: Extensive CArdioVAscular Characterization and Follow-up of Patients Receiving Immune Checkpoint Inhibitors
Acronym: CAVACI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to negative preliminary analysis, slow recruitment (105 patients over 2,5 years), lack of funding, need for more centers, and the changing treatment landscape (approval of ICIs in combination with other cancer treatments).
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christof Vulsteke, Head of Integrated Cancer Center Ghent, Algemeen Ziekenhuis Maria Middelares
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MMS.2021.058
Record Dates: First submitted 2022-12-09; First posted 2023-01-26 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Immune-related Adverse Event; Cardiac Abnormalities, Variable; Immune Checkpoint Inhibitor-Related Myocarditis; Diastolic Dysfunction; Atherosclerosis; Cardiotoxicity
Keywords: Cardio-oncology; Immune-related adverse event; Immune checkpoint inhibitor; Myocarditis; Troponin
MeSH Terms: conditions — Neoplasms; Atherosclerosis; Cardiotoxicity; Myocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cancer patients with a solid tumour eligible for treatment with immune checkpoint inhibitors (Other): Patients are treated as standard of care
  Interventions: Procedure: Cardiology consultation; Diagnostic Test: Chest Computed Tomography (CT) without contrast; Procedure: Non-invasive endothelial function tests; Procedure: Electrocardiogram; Diagnostic Test: Extra serum sample (7.5 mL)

INTERVENTIONS:
Procedure: Cardiology consultation — * Electrocardiogram (ECG).
  * Echocardiogram: A comprehensive evaluation of systolic and diastolic function, ventricular and atrial geometry will be performed. Special attention will be given to acquire a 3D measurement of left ventricular ejection fraction (LVEF) and to perform deformation imaging of left ventricle (global longitudinal strain (GLS)). The right ventricular function will be evaluated by tricuspid annular plane systolic excursion (TAPSE) and peak systolic velocity S' derived from color coded tissue Doppler imaging (TDI). Diastolic dysfunction will be based on average E/e' ratio > 15 and left atrial (LA) area > 30 cm2.
Diagnostic Test: Chest Computed Tomography (CT) without contrast — Calcium score. This will be performed at baseline, 12 and 24 months. The scans at 12 and 24 months will be combined, if possible, with standard of care scans for cancer treatment.
  Other Names: Cardiac CT
Procedure: Non-invasive endothelial function tests — * FMD
  * PAT
  This aspect of the study will only be performed in the patients included by the Antwerp University Hospital due to organizational/practical issues.
  Other Names: Flow mediated dilatation (FMD); Peripheral arterial tonometry (PAT)
Procedure: Electrocardiogram — An ECG will be taken prior to each ICI cycle during the first three months of treatment.
  Other Names: ECG
Diagnostic Test: Extra serum sample (7.5 mL) — An extra serum sample will be taken at baseline, 3, 6, 12, 24 months and in case of sudden cardiac problems. This will subsequently be analysed to determine high-sensitivity troponin I, high-sensitivity troponin T and NT-proBNP.

SUMMARY:
The goal of this prospective, multicentre study is to investigate short- and long-term cardiovascular effects in cancer patients treated with immune checkpoint inhibitors (ICIs).

The main question[s] it aims to answer are:

* To investigate troponin and NT-proBNP values in patients receiving ICIs and their association with ICI-induced CV abnormalities and MACEs.
* Study the calcium score, systolic, and diastolic (dys)function.
* Evaluate associations between patient/disease characteristics / transthoracic echocardiography parameters / electrocardiography parameters and troponin / NT-proBNP levels.

Participants will be closely monitored by performing the following additional visits and testing:

* Chest CT scan prior to treatment start, after 12 and 24 months.
* Consultation with a cardiologist at baseline, 3, 6, 12 and 24 months, who will perform an electrocardiogram and echocardiogram.
* One additional blood sample prior to treatment start, after 3, 6, 12 and 24 months. An extra blood sample could be taken in case of sudden heart problems.
* Non-invasive endothelial function tests prior to treatment start, after 12 and 24 months.

DETAILED DESCRIPTION:
The increasing use of immune checkpoint inhibitors (ICIs) in the treatment of both advanced and early stages of various malignancies has resulted in a substantial increase in the incidence of cardiovascular immune related adverse events (irAEs). The current guidelines are based on anecdotal evidence and expert opinions due to the lack of solid data and prospective studies. Therefore, cardiac monitoring, in patients receiving ICIs, is often not implemented by oncologists as many questions remain unanswered. Hence, the urgent need to investigate the possible short and long term cardiovascular effects of ICIs.

The investigators developed a multicentre, prospective study in which patients with a solid tumour eligible for ICI treatment will be enrolled. The study exists of routine investigations of blood parameters (troponin and (N-terminal) brain-type natriuretic peptide levels in particular) and a thorough cardiovascular follow-up on fixed time points during a period of two years. The cardiovascular follow-up consists of continuous remote patient monitoring, routine cardiology consultations including electrocardiograms, transthoracic echocardiograms, CT-scans for calcium scoring and non-invasive endothelial function tests. Associations between these blood parameters and short and long term cardiovascular irAEs will be statistically analysed.

This project will allow for a better estimate of the incidence of both short and long-term cardiovascular irAEs in a 'real world' patient population receiving ICIs. If the investigators are able to accurately predict and detect short- and long-term cardiovascular irAEs in an early (and subclinical) stage by correct implementation and interpretation of existing cardiac markers, they could be managed early on in a more effective manner.

ELIGIBILITY:
Inclusion Criteria:

* Have a solid tumour and will receive one of the following therapies based on current evidence based clinical guidelines: anti-programmed cell death protein-1 (PD-1), anti-programmed cell death ligand-1 (PD-L1) and/or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) therapy
* Be literate in Dutch or English

Exclusion Criteria:

* Prior treatment with immunotherapy (immune checkpoint inhibitors, T-cell transfer therapy, cancer treatment vaccines or immune system modulators).
* Patients who will receive ICIs in combination with an additional systemic anti-cancer regimen (chemotherapy, tyrosine kinase inhibitors,…).
* Having a known history of human immunodeficiency virus (HIV) infection.
* Having a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as detectable RNA via qualitative nucleic acid testing) infection.
* Having a diagnosis of immunodeficiency or is receiving chronic/active systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
The incidence of an elevated hs-TnT above the ULN if the baseline value was normal; or 1.5 ≥ times baseline if the baseline value was above the ULN within the first three months of treatment. The maximum measured value will be taken into account. | Preliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and 3 months after last patient is included.
  For the primary endpoint, the cumulative incidence of troponin elevation will be calculated with death as a competing risk. Cumulative incidences and corresponding 95% confidence intervals will be reported and a cumulative incidence plot will be used to visualize the results.

SECONDARY OUTCOMES:
The incidence of hs-TnT/NT-proBNP elevations at 6, 12, and 24 months. | Through study completion, an average of 1 year
  Cumulative incidences and 95% confidence intervals, considering death as a competing event.
The incidence of hs-TnT/NT-proBNP elevations at baseline, 3, 6, 12, and 24 months. | Preliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and through study completion, an average of 1 year
  Cumulative incidences and 95% confidence intervals, considering death as a competing event.
Evolution of hs-TnT/NT-proBNP in 24 months compared to baseline. | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual.
Evolution of transthoracic 3D echocardiography parameters (dimensions, diastolic function, valvular abnormalities, LVEF, strain analysis) at baseline, 3, 6, 12, and 24 months. | reliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual.
Evolution of electrocardiography parameters (rhythm, heart axis, PQ interval, QRS duration, bundle branch block, QT interval, RR interval, pathological Q's, left ventricular hypertrophy and STT segments) at baseline, 3, 6, 12, and 24 months. | reliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual.
Association between the evolution of troponin/NT-proBNP and transthoracic echocardiography parameters at baseline, 3, 6, 12, and 24 months. | reliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual.
Association between the evolution of troponin/NT-proBNP and electrocardiography (rhythm, heart axis, PQ, QRS, bundle branch block, QT, RR, pathological Q's, left ventricular hypertrophy and STT segments) parameters at baseline, 3, 6, 12, and 24 months. | reliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual.
Cumulative incidence of cardiovascular (CV) abnormalities at 3, 6, 12, and 24 months based on the CARDIOTOX classification system of Sendón et al., with the inclusion of pericardial effusion and new arrhythmias. | Through study completion, an average of 1 year
  Cumulative incidences and 95% confidence intervals, considering death as a competing event.
Association between the evolution of troponin/NT-proBNP and CV abnormalities (as classified based on the CARDIOTOX classification for myocardial injury including cardiac biomarkers, symptoms, LVEF, LA area, LVESV, GLS and diastolic function). | Through study completion, an average of 1 year
  Joint model combining a linear mixed model for troponin and a sub-distributional proportional hazards model for the time-to-event taking into account death as a competing event for CV abnormality and MACE.
Cumulative incidence of MACEs at 3, 6, 12, and 24 months. MACEs were defined as the composite outcome of nonfatal stroke, nonfatal myocardial infarction, hospital admission for heart failure (HF) and cardiac revascularization, and CV death. | Through study completion, an average of 1 year
  Cumulative incidences and 95% confidence intervals, considering death as a competing event.
Overall survival. | reliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and through study completion, an average of 1 year
  Cumulative incidences and 95% confidence intervals
Association between the evolution of troponin/NT-proBNP and MACEs over a period of two years. Nonfatal stroke, nonfatal myocardial infarction, hospital admission for heart failure, cardiac revascularization and CV death will be combined to report MACEs. | Through study completion, an average of 1 year
  Joint model combining a linear mixed model for troponin and a sub-distributional proportional hazards model for the time-to-event taking into account death as a competing event for CV abnormality and MACE.
The difference in the evolution of hs-TnT/NT-proBNP between combination therapy and monotherapy over a period of two years. | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual. This model will be extended with patient and treatment characteristics and their interaction with time, to evaluate their impact on the evolution of these parameters.
The difference in the evolution of transthoracic echocardiography parameters (dimensions, diastolic function, valvular abnormalities, LVEF, strain analysis) between combination therapy and monotherapy over a period of two years. | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual. This model will be extended with patient and treatment characteristics and their interaction with time, to evaluate their impact on the evolution of these parameters.
The difference in the evolution of electrocardiography parameters (rhythm, heart axis, PQ, QRS, bundle branch block, QT, RR, pathological Q's, left ventricular hypertrophy and STT segments) between combination therapy and monotherapy. | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual. This model will be extended with patient and treatment characteristics and their interaction with time, to evaluate their impact on the evolution of these parameters.
Association between patient characteristics (demographics, medical history, current oncological disease, prior cancer history, prior/concomitant medication and other relevant parameters) and troponin. | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual. This model will be extended with patient and treatment characteristics and their interaction with time, to evaluate their impact on the evolution of these parameters.
Association between patient characteristics (demographics, medical history, current oncological disease, prior cancer history, prior/concomitant medication and other relevant parameters) and NT-proBNP. | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual. This model will be extended with patient and treatment characteristics and their interaction with time, to evaluate their impact on the evolution of these parameters.
Agreement between hs-TnT and hs-TnI levels at baseline, 3, 6, 12, and 24 months. | reliminary analysis once 50 patients have reached their 3-month cardiac follow-up visit and through study completion, an average of 1 year
  Bland-Altman curves and intraclass correlation coefficient (ICC) based on a two-way mixed effects model. The ICC and 95% confidence interval will be reported.
The proportion of severe immune-related non-CV toxicities (grades 3-5). | Through study completion, an average of 1 year
  Proportions and 95% confidence interval
Association between the evolution of troponin/NT-proBNP and severe immune-related non-CV toxicities (grades 3-5, e.g. pneumonitis, colitis, thyroiditis, etc. according to the CTCAE criteria). | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual. This model will be extended with patient and treatment characteristics and their interaction with time, to evaluate their impact on the evolution of these parameters.
Association between the evolution of troponin/NT-proBNP and overall survival. | Through study completion, an average of 1 year
  Joint model combining a linear mixed model for troponin and a sub-distributional proportional hazards model for the time-to-event taking into account death as a competing event for CV abnormality and MACE.
Association between the evolution of troponin and diastolic function (based on the recommendations listed in https://doi.org/10.1016/j.echo.2016.01.011, mitral inflow, tissue doppler imaging parameters). | Through study completion, an average of 1 year
  Linear mixed effects model with a random intercept per subject to account for the correlation measurements coming from the same individual. This model will be extended with patient and treatment characteristics and their interaction with time, to evaluate their impact on the evolution of these parameters.
Calcium score at baseline, 12 months, and 24 months. | Through study completion, an average of 1 year
  Proportions and 95% confidence interval
Peripheral vascular function at baseline, 3 months, 6 months, 12 months and 24 months. | Through study completion, an average of 1 year
  Flow mediated dilatation: dilatation % from baseline to maximal post-occlusion diameter.
  Peripheral arterial tonometry ratio: based on the response to reactive hyperemia using post and pre-occlusion values
Association between the evolution of troponin and calcium score. | Through study completion, an average of 1 year
  Flow mediated dilatation: dilatation % from baseline to maximal post-occlusion diameter.
  Peripheral arterial tonometry ratio: based on the response to reactive hyperemia using post and pre-occlusion values

CONTACTS AND LOCATIONS:
Overall Officials: Christof Vulsteke, Prof, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (4):
- Belgium (4):
  - Antwerp University Hospital, Antwerp, Antwerp
  - AZ Sint-Vincentius Deinze, Deinze, East-Flanders
  - Algemeen Ziekenhuis Maria Middelares, Ghent, East-Flanders
  - AZ Sint-Elisabeth Zottegem, Zottegem, East-Flanders

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delombaerde D, De Sutter J, Croes L, Vervloet D, Moerman V, Van de Veire N, Willems AM, Wouters K, Peeters M, Prenen H, Vulsteke C. Extensive CArdioVAscular Characterization and Follow-Up of Patients Receiving Immune Checkpoint Inhibitors: A Prospective Multicenter Study. Pharmaceuticals (Basel). 2023 Apr 20;16(4):625. doi: 10.3390/ph16040625. PMID 37111382